CLINICAL TRIAL: NCT02263781
Title: PREPL in Health and Disease
Acronym: PHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S57206
Record Dates: First submitted 2014-10-01; First posted 2014-10-13 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Hypotonia-Cystinuria Syndrome; Muscle Hypotonia; Healthy Volunteers; Dwarfism, Growth Hormone Deficiency; Obesity; Prader-Willi Syndrome
MeSH Terms: conditions — Hypotonia-Cystinuria Syndrome; Muscle Hypotonia; Dwarfism, Pituitary; Obesity; Prader-Willi Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control Blood (Experimental): Patients on routine postinfectious control, blood draw
  Interventions: Procedure: Blood draw
- Primary PREPL deficiency Blood (Experimental): Patients with primary PREPL deficiency, blood draw
  Interventions: Procedure: Blood draw
- Prader Willi syndrome Blood (Experimental): Patients with Prader-Willi syndrome, blood draw
  Interventions: Procedure: Blood draw
- Primary PREPL deficiency like Blood (Experimental): Patients with symptoms overlapping with primary PREPL deficiency (like hypotonia, growth hormone deficiency, obesity), blood draw
  Interventions: Procedure: Blood draw
- Control muscle (Experimental): Patients without hypotonia, growth hormone deficiency, obesity, undergoing elective surgery, muscle biopsy from the surgical site and blood draw
  Interventions: Procedure: Blood draw; Procedure: muscle biopsy
- Prader-Willli syndrome muscle (Experimental): Patients with Prader-Willi syndrome undergoing elective anesthesia or surgery, muscle biopsy (from surgical site if applicable) and blood draw
  Interventions: Procedure: Blood draw; Procedure: muscle biopsy

INTERVENTIONS:
Procedure: Blood draw — Blood draw
Procedure: muscle biopsy — Muscle biopsy during planned anesthesia/surgery
  Arms: Control muscle; Prader-Willli syndrome muscle

SUMMARY:
Evaluation of PREPL activity in healthy controls and known or possible PREPL deficient patients

DETAILED DESCRIPTION:
PREPL is defective in hypotonia cystinuria syndrome and in isolated PREPL deficiency. The investigators have constructed a blood test to evaluate PREPL activity in patients with possible PREPL deficiency.

The study will determine normal values for age (0-18) for PREPL activity in blood.

Also, patients with a clinical phenotype that overlaps with PREPL deficiency (including patients with known primary PREPL deficiency and Prader-Willi syndrome) will be evaluated for PREPL activity in blood.

A last part of the study will involve muscle biopsies during elective anesthesia/surgery for other reasons. There will be 2 groups: patients without signs of PREPL deficiency undergoing surgery (controls) and patients with Prader-Willi syndrome undergoing anesthesia or surgery (patients). The control group will be age-matched to the hypotonia group. In the muscle biopsies, PREPL activity and expression will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* According to group
* Control group: children seen at a postinfectious consultation

Exclusion Criteria:

* Control group: symptoms overlapping with PREPL deficiency, genetic or syndromic disease, atypically developing children
* other groups: contraindication for blood draw
* group with muscle biopsy: contra-indication for muscle biopsy

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2014-10; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
PREPL activity (ng active PREPL/g protein) normal values in blood | 3 months
  normal values for PREPL activity
PREPL activity in patients with Prader Willi syndrome compared to activity in normal controls | 3 months
  Comparison of PREPL activity in blood and muscle between above mentioned groups
PREPL activity in patients with primary PREPL deficiency compared to activity in normal controls | 3 months
  Comparison of PREPL activity in blood between above mentioned groups

SECONDARY OUTCOMES:
PREPL activity in patients with muscle weakness/obesity/growth hormone deficiency compared to activity in normal controls | 3 months
  exploratory evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Luc Régal, MD, Principal Investigator — KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

REFERENCES:
- [Background] Regal L, Shen XM, Selcen D, Verhille C, Meulemans S, Creemers JW, Engel AG. PREPL deficiency with or without cystinuria causes a novel myasthenic syndrome. Neurology. 2014 Apr 8;82(14):1254-60. doi: 10.1212/WNL.0000000000000295. Epub 2014 Mar 7. PMID 24610330
- [Background] Jaeken J, Martens K, Francois I, Eyskens F, Lecointre C, Derua R, Meulemans S, Slootstra JW, Waelkens E, de Zegher F, Creemers JW, Matthijs G. Deletion of PREPL, a gene encoding a putative serine oligopeptidase, in patients with hypotonia-cystinuria syndrome. Am J Hum Genet. 2006 Jan;78(1):38-51. doi: 10.1086/498852. Epub 2005 Nov 23. PMID 16385448